CLINICAL TRIAL: NCT04657237
Title: Effect of Anesthesia and Surgical Stress on the Expression of Programmed Death-1 and Programmed Death-1 Ligand on T Lymphocyte After Breast Cancer Surgeries
Brief Title: Effect of Anesthesia on Expression of Programmed Death-1 and Programmed Death-1 Ligand in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lecturer of anesthesia, ICU and pain managment, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 359
Record Dates: First submitted 2020-11-17; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Programmed Cell Death 1
Keywords: brest cancer; programmed cell death1; programmed cell death ligand 1

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): all patients will receive general anesthesia and will receive intravenous paracetamol (1 g) before skin closure and then given every 6 hrs in the 1st postoperative day
- TPVB group (Active Comparator): Patients will receive total volume (20 ml) 0.25% bubivicaine divided equally at each level of T4 and T6 at thoracic paravertebral space then they will recive general anesthesia.
  Interventions: Procedure: Thoracic Paravertebral block

INTERVENTIONS:
Procedure: Thoracic Paravertebral block — TPVB will be given using high frequency linear U/S transducer, place the U/S ultrasound probe was placed parallel to the vertebral spine at T4, and, T6 level and shifted 2-3 cm laterally to obtain the appropriate visualization. Following the identification of pleura, transverse process and paravertebral space, the needle was inserted in caudocranial direction using in-plane approach. Confirm negative vessel or pleural breach via aspiration then proceed with local anaesthetic 0.25% bupivacaine (20 ml) delivery slowly divided equally at T4and T6; the pleura will be seen to be pushed downward
  Arms: TPVB group

SUMMARY:
Surgery is first-line treatment for solid tumors. However, surgical trauma-induced physiologic stress has been demonstrated to facilitate metastasis and recurrence in different types of cancer. It has been reported that the PD-1/PD-L1 pathway could be activated by surgical stress. Hence, we instigate the effect of anesthetic technique on expression of PD1 and PD1 ligand.

DETAILED DESCRIPTION:
The cellular immune response plays a central part in postoperative clearance of tumor cells. T lymphocytes and natural killer (NK) cells are two predominant cytotoxic effector cells that are the major components of antitumor immunity. In mouse models, proliferation of T lymphocytes in response to surgical trauma is defective . Programmed death-1 (PD-1) belongs to the CD28 receptor superfamily. It is an inhibitory receptor, and its expression is upregulated on activated leukocytes, resulting in an inhibited immune response. PD-1 interacts with two ligands: programmed death ligand-1 (PD-L1, also referred to as B7-H1) and programmed death ligand-2 (PD-L2, also known as B7-DC). PD-L2 is expressed mainly on activated dendritic cells (DCs) and macrophages, whereas PD-L1 is distributed widely. In addition to immune cells, some subsets of tumor cells also express PD-L1 to escape from immunosurveillance. It has been reported that the PD-1/PD-L1 pathway could be activated by surgical stress. Hence, we instigate the effect of anesthetic technique on expression of PD1 and PD1 ligand.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for breast cancer surgery

Exclusion Criteria:

* compromised immune function (such as infection with the human immunodeficiency virus, immunodeficiency, or treatment with corticosteroids, immunosuppressive drugs, or chemotherapy)
* ASA > III
* age> 70 years old.
* patients refusal to the procedure.
* Infection of the skin at or near site of needle puncture.
* Coagulopathy .
* Drug hypersensitivity or allergy to the studied drugs.
* Central or peripheral neuropthy .
* Pre-operative opoid consumption ( within 24 hours preoperative )
* Anomalies of the vertebral column .

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
change in level of PD1 and PD1 ligand postoperatively | preoerative (day-0),1st day, and 3 rd day after surgery
  blood sample will be withdrawn and human peripheral blood monocyte cells (PBMCs) will be separated with a Ficoll-Isopaque density gradient. Flow cytometric analyses will be carried out immediately. For ex vivo experiments, PBMCs will be cultured with Iscove's modified Dulbecco's medium (IMDM) containing 10 % human serum albumin.

SECONDARY OUTCOMES:
total request of analgesia | 24 hours postoperative
  the total amount of analgesia (paracetamol) will be recorded and calculated

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No